CLINICAL TRIAL: NCT04351841
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Investigate the Effect of an Arabinogalactan Product for 6 Weeks on the Gut Microbiome in Adults
Brief Title: To Investigate the Effect of Arabinogalactan on the Gut Microbiome in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biofortis, Merieux NutriSciences (Industry)
Collaborators: Lonza Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO 1906
Record Dates: First submitted 2020-04-07; First posted 2020-04-17 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Gut Microbiota
Keywords: microbiome; stool; indigestible carbohydrate
MeSH Terms: interventions — arabinogalactan; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): 15 g maltodextrin per day consumed in the morning
  Interventions: Other: maltodextrin
- Active (Experimental): 15 g arabinogalactan per day consumed in the morning
  Interventions: Other: arabinogalactan

INTERVENTIONS:
Other: arabinogalactan — A beverage will be prepared by thoroughly mixing the 15 g of arabinogalactan with water and Crystal Light flavoring
  Arms: Active
Other: maltodextrin — A beverage will be prepared by thoroughly mixing the 15 g of maltodextrin with water and Crystal Light flavoring
  Arms: control

SUMMARY:
Dietary fiber is an important nutrient that supports gastrointestinal function, as well as the maintenance of blood glucose and cholesterol. Additionally, it is suggested that dietary fiber may provide other health benefits, such as maintenance of healthy weight through effects on satiety. Furthermore, dietary fiber can improve health by modulating the microbial communities residing in human gut, particularly in the large intestine. The microbes in the gut modulate a wide variety of biological processes essential for health of the host. Currently, the average intake of fiber in the U.S. is ~40-50% below adequate intake levels.

ResitAid, a Lonza's arabinogalactan, is a hemicellulose that is abundant in plants. Arabinogalactans including ResitAid are found in seeds, leaves, roots, and fruit of higher plants, such as cereals, beans, leeks, pear, corn, bark, and wheat. ResitAid, the arabinogalactan ingredient used in this study, is isolated from larch (Larix laricina) using a patented water-based extraction process. ResitAid has been designated as Generally Recognized as Safe (GRAS) by the U.S. FDA for multiple uses and has been used in numerous previous clinical studies in humans, with no significant safety issues observed at intakes of up to 30 g daily for up to 6 weeks. It was reported that 15 g and 30 g of different preparation of arabinogalactan could significantly increase certain microbial populations considered to be beneficial (e.g., Lactobacillus spp.). Nevertheless, more clinical evidence is needed to support the effect of ResistAid on the microbial composition in the gut. This study is designed to investigate the effect of daily consumption of 15 g of ResitAid on the gastrointestinal microbial profile and fecal short-chain fatty acid contents in healthy adults.

Primary Objective: Modulation of the microbiome

Secondary objectives:

1. Changes in Lactobacillus ssp.
2. Changes in Bifidobacterium ssp.
3. Changes in SCFA
4. Changes in bowel movement
5. Changes in the SF-36 questionnaire

DETAILED DESCRIPTION:
The study is a randomized, crossover, single-center trial with one screening visit (Visit 1; Week -1) and 2 test periods [Test Period I (Visits 2, 3, and 4; Weeks 0, 3, and 6) and Test Period II (Visits 5, 6, and 7; Weeks 9, 12 and 15)] separated by a minimum 3-week washout period.

At Visit 1 (Week -1), subjects will provide informed consent and undergo assessments of medical history and medication/supplement use, and inclusion and exclusion criteria. Fasting (12 ± 2 h) blood samples will be collected for chemistry and hematology. Subjects will be counseled to exclude fermented foods or beverages that do or might contain live probiotics (e.g., yogurt, kombucha). Subjects will also be dispensed a gastrointestinal (GI) and Bowel Habits Diary and stool collection kit. Subjects will be instructed to complete the GI and Bowel Habits Diary during the 3 days prior to Visit 2 (Week 0) and to collect fecal samples from one bowel movement during the 3 days prior to Visit 2 (Week 0).

At Visit 2 (Week 0), subjects will arrive at the clinic fasted (12 ± 2 h, water only) to undergo clinic visit procedures. Adverse events (AE) will be assessed and the SF-36 Questionnaire will be administered. Fecal samples will be collected and the GI and Bowel Habits Diary will be collected and reviewed. Subjects will be randomly assigned to a study product for home consumption with or without breakfast in the morning. Subjects will be dispensed a GI and Bowel Habits Diary and stool collection kit and will be instructed to complete the diary during the 3 days immediately prior to Visit 3 (Week 3) and to collect fecal samples from one bowel movement during the same 3 days immediately prior to Visit 3 (Week 3).

At Visit 3 (Week 3), subjects will return to the clinic for clinic visit procedures. AEs will be assessed and the SF-36 Questionnaire will be administered. The fecal samples will be collected and the GI and Bowel Habits Diary will be collected and reviewed. Study product will be re-dispensed back to subjects for home consumption. Subjects will be dispensed a GI and Bowel Habits Diary and stool collection kit and will be instructed to complete the diary during the 3 days immediately prior to Visit 4 (Week 6) and to collect fecal samples during the same period.

At Visit 4 (Week 6), subjects will arrive at the clinic fasted (12 ± 2 h, water only) to undergo clinic visit procedures. AEs will be assessed and the SF-36 Questionnaire will be administered. Subjects will be queried about compliance with study instructions. The fecal samples will be collected and GI and Bowel Habits Diary will be collected and reviewed. Fasting (12 ± 2 h) blood samples will be collected for chemistry and hematology. Subjects will be dispensed a stool collection kit and will be instructed to collect fecal samples from one bowel movement during the 3 days immediately prior to Visit 5 (Week 9). Subjects will be instructed to begin the 3-week washout period and return to the clinic to begin Test Period II at Visit 5 (Week 9).

At Visit 5 (Week 9), subjects will return to the clinic fasted (12 ± 2 h, water only), crossover to the other study product in their test sequence, and repeat the procedures from Visits 2 (Week 0) with the exclusion of the randomization procedure. At Visit 6 (Week 12), subjects will repeat the procedures from Visit 3 (Week 3) and at Visit 7 (Week 15), subjects will repeat the procedures from Visit 4 (Week 6). Subjects will be dismissed at the end of Visit 7.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 18.0 to 32.0 kg/m2, inclusive, at Visit 1 (Week -1).
2. Self-reported regular bowel movement at Visit 1 (Week -1).
3. Non-user of all tobacco and smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes) and nicotine products (e.g., nicotine patches, nicotine gums) and has no plans to change smoking habits during the study period.
4. Non-user of any marijuana or hemp products and has no plans to use marijuana or hemp products during the study period.
5. Willing to maintain physical activity patterns, body weight, and habitual diet throughout the trial, except for exclusion of fermented foods that do or might contain live probiotics (e.g., yogurt, kombucha) and inclusion of study products.
6. Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to and during Visits 1, 2, 4, 5, and 7 (Weeks -1, 0, 6, 9, and 15).
7. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
8. Willing and able to comply with the visit schedule and fecal sample collection/processing/storage requirements during the study period.
9. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
10. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Abnormal laboratory test results of clinical significance at Visit 1 (Week -1), at the discretion of the Clinical Investigator. One re-test will be allowed on a separate day prior to Visit 2 (Week 0), for subjects with abnormal laboratory test results.
2. Clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, gastric reflux, indigestion, dyspepsia, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose and gluten intolerance or allergies).
3. Recent (within 2 weeks of Visit 1; Week -1) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as ≥3 loose or liquid stools/day).
4. Self-reported history (within 6 weeks of Visit 1; Week -1) of constipation (defined as <3 bowel movements per week).
5. History or presence of uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine, hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders.
6. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Week -1).

   One re-test will be allowed on a separate day prior to Visit 2 (Week 0), for subjects whose blood pressure exceeds either of these cut points at Visit 1 (Week -1), in the judgment of the Clinical Investigator.
7. Known allergy intolerances or sensitivity to any of the ingredients in the study product (Appendix 8).
8. Extreme dietary habits (e.g., Atkins diet/ketogenic diet, very high protein, very high fiber, vegetarian), in the opinion of the Clinical Investigator.
9. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
10. Major trauma or any other surgical event within 3 months of Visit 1 (Week -1).
11. Signs or symptoms of an active infection of clinical relevance within 5 days of Visit 1 (Week -1). The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to Visit 1 (Week -1). If an infection occurs during the study period, test visits will be rescheduled until all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to study visits.
12. Weight loss or gain >4.5 kg in the 3 months prior to Visit 1 (Week -1).
13. Currently or planning to be on a weight loss regimen during the duration of the study.
14. Antibiotic use within 2 months of Visit 1 (Week -1).
15. Use of steroids within 1 month of Visit 1 (Week -1).
16. Chronic use (i.e., daily on a regular basis) of anti-inflammatory medications (e.g., NSAIDs) within 1 month of Visit 1 (Week -1).
17. Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to prebiotics or probiotics, laxatives, enemas, fiber supplements and/or suppositories, anti-diarrheal agents, and/or anti-spasmodic within 2 weeks of Visit 1 (Week -1).
18. Bismuth subsalicylate (e.g., Pepto Bismol) and antacids (e.g., Tums) ≤2 times/ week starting from 2 weeks prior to Visit 1 (Week -1), with the exception of 7 days prior to the stool collection period, during which consumption of these products are not allowed.
19. Consumption of fermented foods or beverages that do or might contain live probiotics (Appendix 1) within 2 weeks of Visit 1 (Week -1).
20. Participated in colonoscopy or colonoscopy preparation within 3 months prior to Visit 1 (day -14).
21. Exposure to any non-registered drug product within 4 weeks prior to Visit 1 (Week - 1).
22. Recent history of (within 12 months of screening; Visit 1; Week -1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
23. Has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
composition of fecal microbiome | up to 6 weeks
  relative abundance of bacteria and alpha- and beta-diversity
Concentration of fecal short-chain fatty acids | Change from the baseline at 6 weeks
  acetate, butyrate, propionate, valerate, isobutyrate, and isovalerate contents (ug/g wet stool)

SECONDARY OUTCOMES:
Bowel Movement | Change from the baseline at 6 weeks
  Number per week
stool consistency | Change from the baseline at 6 weeks
  Using Bristol Stool Scale [ranging from 1 (solid, hard) to 7 (losse)] to assess stool consistency for 7 days
sensation of incomplete evacuation during bowel movement | Change from the baseline at 6 weeks
  self-assess for 7 days using a Likert 4-point scale
straining during bowel movement | Change from the baseline at 6 weeks
  self-assess for 7 days using a Likert 4-point scale
discomfort during bowel movement | Change from the baseline at 6 weeks
  self-assess for 7 days using a Likert 4-point scale
general health status | Change from the baseline at 6 weeks
  SF-36 questionnaire measures general health status and health-related quality of life. The score ranges from 0 to 100 with the highest value indicating a favorable health state.
Concentration of plasma short-chain fatty acids | Change from the baseline at 6 weeks
  acetate, butyrate, propionate, valerate, isobutyrate, and isovalerate contents (umol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Oliver Chen, Addison, Illinois, United States